CLINICAL TRIAL: NCT03121365
Title: Digital Literacy Promotion Among Medicaid Children
Brief Title: Digital Literacy Promotion
Acronym: DLP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Vanguard Strong Start for Kids Program (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 16-013524
Record Dates: First submitted 2017-04-17; First posted 2017-04-20 (Actual); Results first posted 2019-11-20 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Language Development; Literacy
Keywords: Digital literacy; Reading
MeSH Terms: conditions — Literacy

STUDY DESIGN:
Intervention Model Description: Eligible participants will be stratified by site and randomized 1:1
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard/Board Book Arm (Active Comparator): Parent-infant dyads randomized to the standard/board book arm will receive developmentally appropriate early reader board books at the time of their infant's 6, 9, and 12 month well visits. In addition to the books, parent-infant dyads will be provided information on the importance of early parent-child reading activity by pediatric clinicians using the Reach Out and Read framework.
  Interventions: Behavioral: Standard/Board Book Arm
- Digital/E-Book Arm (Experimental): Parent-infant dyads randomized to the digital/e-book arm will receive developmentally appropriate e-books at the time of their infant's 6, 9, and 12 month well visits. In addition to the books, parent-infant dyads will be provided information on the importance of early parent-child reading activity by pediatric clinicians using the Reach Out and Read framework.
  Interventions: Behavioral: Digital/E-Book Arm

INTERVENTIONS:
Behavioral: Digital/E-Book Arm — Promotion of early reader digital e-book reading
  Arms: Digital/E-Book Arm
Behavioral: Standard/Board Book Arm — Promotion of early reader board book reading
  Arms: Standard/Board Book Arm

SUMMARY:
This study evaluates the effects of digital versus standard literacy promotion, as well as dialogic language behaviors and reading comprehension among infants when comparing the use of e-books to standard board books. Around half of the participants will receive standard board books at the 6, 9, and 12 month well visits, while the other half will receive digital e-books.

DETAILED DESCRIPTION:
This study has three main objectives. The first is to test the effects of digital versus standard literacy promotion by way of a randomized controlled trial design. The second aim is to explore the reading behaviors and reading activities between parents and their infants when comparing the use of e-books to standard board books. The third aim is to identify themes regarding dialogical reading behaviors among parents participating in the video sub-study.

Participants will be stratified by clinic site and randomized to receive literacy promotion using 1) standard early reader board books or 2) digital electronic early reader e-books. We will recruit and consent one hundred eligible parent-infant dyads, with the infant being between 5 and 7 months of age at enrollment.

In this intervention, parent-infant dyads randomized to the digital arm will receive developmentally appropriate e-books. Those randomized to the standard arm will receive developmentally appropriate board books. Participants will receive either the e-book or board book at the time of their 6, 9 and 12 month well visits. In addition to the books, parent-infant dyads in both arms will be provided information on the importance of early parent-child reading activity by pediatric clinicians using the Reach Out and Read framework.

The main outcome will be differences in Bayley-3 Composite scores between groups. Secondary aims include differences in StimQ Reading Subscale Scores and Edinburgh Postnatal Depression Scale Scores between groups.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking
* Parents ≥ 15 years of age at start of study
* Child born ≥ 35 weeks estimated gestational age
* Child 5 to 7 months
* Medicaid Insurance
* Access to a smart phone and/or tablet

Exclusion Criteria:

* Child has neurodevelopmental disabilities or congenital malformation

Ages: 5 Months to 7 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Guevara, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Following completion of all analyses, data will be de-identified and made available for other investigators.
Supporting Information: Study Protocol
Time Frame: 12 months after publication of all relevant papers
Access Criteria: De-identified only

REFERENCES:
- [Derived] Guevara JP, Erkoboni D, Gerdes M, Winston S, Sands D, Rogers K, Haecker T, Jimenez ME, Mendelsohn AL. Promoting Early Literacy Using Digital Devices: A Pilot Randomized Controlled Trial. Acad Pediatr. 2021 Aug;21(6):1001-1008. doi: 10.1016/j.acap.2021.05.013. Epub 2021 May 19. PMID 34022425

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard/Board Book Arm: Parent-infant dyads randomized to the standard/board book arm will receive developmentally appropriate early reader board books at the time of their infant's 6, 9, and 12 month well visits. In addition to the books, parent-infant dyads will be provided information on the importance of early parent-child reading activity by pediatric clinicians using the Reach Out and Read framework.
  Standard/Board books: Promotion of early reader board book reading
- Digital/E-Book Arm: Parent-infant dyads randomized to the digital/e-book arm will receive developmentally appropriate e-books at the time of their infant's 6, 9, and 12 month well visits. In addition to the books, parent-infant dyads will be provided information on the importance of early parent-child reading activity by pediatric clinicians using the Reach Out and Read framework.
  Digital/E-books: Promotion of early reader digital e-book reading
Period: Baseline
Arm/Group | Standard/Board Book Arm | Digital/E-Book Arm
Started | 55 | 49
Completed | 54 | 48
Not Completed | 1 | 1
Period: 1 Months
Arm/Group | Standard/Board Book Arm | Digital/E-Book Arm
Started | 54 | 48
Completed | 52 | 45
Not Completed | 2 | 3
Period: 4 Months
Arm/Group | Standard/Board Book Arm | Digital/E-Book Arm
Started | 54 | 45
Completed | 51 | 44
Not Completed | 3 | 1
Period: 7 Months
Arm/Group | Standard/Board Book Arm | Digital/E-Book Arm
Started | 54 | 45
Completed | 44 | 37
Not Completed | 10 | 8

BASELINE CHARACTERISTICS:
Population: Of the 104 enrolled, 102 were randomized to either study arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard/Board Book Arm | Digital/E-Book Arm | Total
Number analyzed (Participants) | 54 | 48 | 102
Age, Continuous [Mean (Standard Deviation); unit: years]
  Mother's Age | 28.0 (5.1) | 29.6 (6.2) | 28.7 (5.7)
  Father's Age | 31.4 (7.9) | 32.3 (6.4) | 32.0 (7.3)
Age, Customized [Mean (Standard Deviation); unit: months]
  Infant Age | 6.1 (0.40) | 6.2 (0.38) | 6.2 (0.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 23 | 52
  Male | 25 | 25 | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 22 | 23 | 45
  Caucasian | 25 | 17 | 42
  Hispanic or Latino | 2 | 3 | 5
  Other | 5 | 5 | 10
Marital Status [Count of Participants; unit: Participants]
  Single/Never Married | 21 | 17 | 38
  Separated/Divorced | 2 | 1 | 3
  Married/Living Together as if Married | 31 | 30 | 61
Level of Education [Count of Participants; unit: Participants]
  Some High School | 1 | 2 | 3
  High School/GED | 13 | 19 | 32
  Some College | 20 | 15 | 35
  College/Post College Degree | 20 | 12 | 32
Annual Household Income [Count of Participants; unit: Participants]
  $0 - $24,999 | 23 | 19 | 42
  $25,000 - $49,999 | 24 | 19 | 43
  $50,000+ | 7 | 9 | 16
Number of Other Adults in the Household [Mean (Standard Deviation); unit: Adults] | 1.2 (0.9) | 1.5 (0.9) | 1.3 (0.9)
Number of Other Children in the Household [Mean (Standard Deviation); unit: Children] | 1.2 (1.0) | 1.0 (1.1) | 1.2 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Bayley Scales of Infant and Toddler Development (Infant is 12-18 Months Old)
Description: Evaluation of the infant's cognitive, language and motor development using the Bayley Scales of Infant and Toddler Development, Third Edition (BSID-III).
  Results were reported as composites of cognitive, language, and motor scores, where data were continuous variables on a scale with a normal distribution of 95%. The composite scores are scaled to a metric with a mean of 100 and a standard deviation of 15, and range from 40-160. A composite score above 77.5 is considered developmentally average and a composite score below 77.5 is considered a developmental concern. Data were described using mean and standard deviation. Significance was considered at a level of 0.05.
Time Frame: Second Study visit (approximately one month after child is age-eligible for 12 month well child visit)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard/Board Book Arm | Digital/E-Book Arm
Number analyzed (Participants) | 43 | 37
score on a scale
  Cognitive Composite Score | 98.8 (10.5) | 99.6 (11.9)
  Language Composite Score | 89.7 (10.3) | 85.7 (11.2)
  Motor Composite Score | 94.8 (9.4) | 97.4 (9.4)
Statistical Analysis 1: Comparison: Standard/Board Book Arm vs Digital/E-Book Arm; Bayley Scales of Infant and Toddler Development Cognitive Composite Scores between infants 12-18 months old in the Standard and Digital Arms; Test type: Equivalence — 0.05; p = .7635, t-test, 2 sided
Statistical Analysis 2: Comparison: Standard/Board Book Arm vs Digital/E-Book Arm; Language Composite Scores between infants 12-18 months old in the Standard and Digital Arms; Test type: Equivalence — 0.05; p = .0996, t-test, 2 sided
Statistical Analysis 3: Comparison: Standard/Board Book Arm vs Digital/E-Book Arm; Gross Motor Composite Scores between infants 12-18 months old in the Standard and Digital Arms; Test type: Equivalence — 0.05; p = .2291, t-test, 2 sided

2. Secondary Outcome: StimQ READ Subscale Change Score
Description: Differences in StimQ READ Subscale scores collected approximately 1 month after the 6, 9, and 12 month well visits.
  Reading activity is measured using the StimQ READ subscale. This contains "yes/no" questions reflecting access to books, frequency of shared reading, and variety of books read in homes of young children, ages 5 to 36 months. The StimQ-Infant READ subscale is for use with infants 5-12 months of age and the StimQ-Toddler READ subscale is used with toddlers 12-36 months of age. The StimQ Infant and Toddler Read Subscales include a point scale for measuring cognitive stimulation resulting from the reading activity. Scores for the StimQ-Infant READ scale range from 0-15 with higher scores (greater number values) reflective of higher reading exposure. Scores for the StimQ-Toddler READ scale range from 0-19 with higher scores (greater number values) reflective of higher reading exposure.
Time Frame: 1 month after the 6, 9, and 12 month well visits
Population: The variation in number analyzed per row is reflective of participants who had incomplete measures at different study time-points which prevented analysis of their [missing] scores since the analysis is a comparison of scores at different study time-points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard/Board Book Arm | Digital/E-Book Arm
Number analyzed (Participants) | 52 | 44
units on a scale
  Difference in StimQ scores at 7 and 10 months: number analyzed (Participants) | 51 | 42
  Difference in StimQ scores at 7 and 10 months | 0.4 (4.9) | 2.9 (5.4)
  Difference in StimQ scores at 10 and 13 months: number analyzed (Participants) | 44 | 36
  Difference in StimQ scores at 10 and 13 months | 3.5 (2.3) | 2.9 (4.5)
  Difference in StimQ scores at 7 and 13 months: number analyzed (Participants) | 44 | 36
  Difference in StimQ scores at 7 and 13 months | 4.3 (3.5) | 4.9 (4.3)
Statistical Analysis 1: Comparison: Standard/Board Book Arm vs Digital/E-Book Arm; StimQ scores between infants 6 months of age and 9 months of age in the board book arm and e-book arm; Test type: Equivalence — 0.05; p = .0180, t-test, 2 sided
Statistical Analysis 2: Comparison: Standard/Board Book Arm vs Digital/E-Book Arm; StimQ scores between infants 9 months of age and 12 months of age in the board book arm and e-book arm; Test type: Equivalence — 0.05; p = .4144, t-test, 2 sided
Statistical Analysis 3: Comparison: Standard/Board Book Arm vs Digital/E-Book Arm; StimQ scores between infants 6 months of age and 12 months of age in the board book arm and e-book arm; Test type: Equivalence — 0.05; p = .4251, t-test, 2 sided

3. Secondary Outcome: Frequency of Parent-Reported Board Book Reading
Description: Frequency of board book reading in the prior two weeks. Parents reported frequency as very often, often, rarely, never. Very often and often categories were combined and rarely and never categories were combined. We report number in each arm who report very often/often.
Time Frame: 1 month
Population: 3 participants in the DLP arm dropped out prior to completion of 1 month study visit.
Measure: Count of Participants; unit: Participants
Groups:
- Digital/E-Book Arm: Parent-infant dyads randomized to the digital/e-book arm will receive developmentally appropriate e-books at the time of enrollment. In addition to the books, parent-infant dyads will be provided information on the importance of early parent-child reading activity by pediatric clinicians using the Reach Out and Read framework at their infant's 6, 9, and 12 month well visits.
  Digital/E-Book Arm: Promotion of early reader digital e-book reading
Arm/Group | Standard/Board Book Arm | Digital/E-Book Arm
Number analyzed (Participants) | 52 | 45
Participants
  Very Often/Often | 35 | 25
  Rarely/Never | 17 | 20
Statistical Analysis 1: Comparison: Standard/Board Book Arm vs Digital/E-Book Arm; Test type: Superiority; p = 0.235, Chi-squared — Difference in Board Book Reading

4. Secondary Outcome: Frequency of E-Book Reading
Description: Frequency of e-book reading in the prior two weeks. Parents reported frequency as very often, often, rarely, never. Very often and often categories were combined and rarely and never categories were combined. We report number in each arm who report very often/often.
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Standard/Board Book Arm | Digital/E-Book Arm
Number analyzed (Participants) | 52 | 45
Participants
  Very Often/Often | 6 | 33
  Rarely/Never | 46 | 12
Statistical Analysis 1: Comparison: Standard/Board Book Arm vs Digital/E-Book Arm; Test type: Superiority; p < 0.001, Chi-squared

5. Secondary Outcome: Frequency of Television Viewing
Description: Frequency of television viewing in the prior two weeks. Parents reported frequency as very often, often, rarely, never. Very often and often categories were combined and rarely and never categories were combined. We report number in each arm who report very often/often.
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Standard/Board Book Arm | Digital/E-Book Arm
Number analyzed (Participants) | 52 | 45
Participants
  Very Often/Often | 17 | 17
  Rarely/Never | 35 | 28
Statistical Analysis 1: Comparison: Standard/Board Book Arm vs Digital/E-Book Arm; Test type: Superiority; p = 0.601, Chi-squared

6. Secondary Outcome: Frequency of Board Book Reading
Description: as for outcome 3
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard/Board Book Arm | Digital/E-Book Arm
Number analyzed (Participants) | 51 | 44
Participants
  Very Often/Often | 33 | 23
  Rarely/Never | 18 | 21
Statistical Analysis 1: Comparison: Standard/Board Book Arm vs Digital/E-Book Arm; Test type: Superiority; p = 0.219, Chi-squared

7. Secondary Outcome: Frequency of E-Book Reading
Description: as for outcome 4
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard/Board Book Arm | Digital/E-Book Arm
Number analyzed (Participants) | 51 | 44
Participants
  Very Often/Often | 7 | 26
  Rarely/Never | 44 | 18
Statistical Analysis 1: Comparison: Standard/Board Book Arm vs Digital/E-Book Arm; Test type: Superiority; p < 0.001, Chi-squared

8. Secondary Outcome: Frequency of Television Viewing
Description: as for outcome 5
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard/Board Book Arm | Digital/E-Book Arm
Number analyzed (Participants) | 51 | 44
Participants
  Very Often/Often | 18 | 18
  Rarely/Never | 33 | 26
Statistical Analysis 1: Comparison: Standard/Board Book Arm vs Digital/E-Book Arm; Test type: Superiority; p = 0.574, Chi-squared

9. Secondary Outcome: Frequency of Board Book Reading
Description: as for outcome 3
Time Frame: 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard/Board Book Arm | Digital/E-Book Arm
Number analyzed (Participants) | 44 | 37
Participants
  Very Often/Often | 31 | 23
  Rarely/Never | 13 | 14
Statistical Analysis 1: Comparison: Standard/Board Book Arm vs Digital/E-Book Arm; Test type: Superiority; p = 0.430, Chi-squared

10. Secondary Outcome: Frequency of E-Book Reading
Description: as for outcome 4
Time Frame: 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard/Board Book Arm | Digital/E-Book Arm
Number analyzed (Participants) | 44 | 37
Participants
  Very Often/Often | 10 | 24
  Rarely/Never | 34 | 13
Statistical Analysis 1: Comparison: Standard/Board Book Arm vs Digital/E-Book Arm; Test type: Superiority; p < 0.001, Chi-squared

11. Secondary Outcome: Frequency of Television Viewing
Description: as for outcome 5
Time Frame: 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard/Board Book Arm | Digital/E-Book Arm
Number analyzed (Participants) | 44 | 37
Participants
  Very Often/Often | 17 | 15
  Rarely/Never | 27 | 22
Statistical Analysis 1: Comparison: Standard/Board Book Arm vs Digital/E-Book Arm; Test type: Superiority; p = 0.861, Chi-squared

12. Post Hoc Outcome: Feasibility of Literacy Promotion
Description: Proportion of participants in each arm who received books and literacy promotion counseling at well visits and completed all study visits.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard/Board Book Arm | Digital/E-Book Arm
Number analyzed (Participants) | 54 | 48
Participants | 44 | 37

ADVERSE EVENTS:
Time Frame: Adverse Events were monitored throughout study completion, approximately 1 year 8 months
Arm/Group | Standard/Board Book Arm | Digital/E-Book Arm
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/49
Other Adverse Events (participants affected / at risk) | 2/55 | 1/49
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard/Board Book Arm (N=55) | Digital/E-Book Arm (N=49)
Breach of Confidentiality (Social circumstances) | 2 (2) | 1 (1)

LIMITATIONS AND CAVEATS:
1. We were not able to control for use of digital devices by participants in the board book arm, which may affect home reading environment outcomes
2. Pilot study and small sample size and small power may affect significance of outcome measures

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-10): https://cdn.clinicaltrials.gov/large-docs/65/NCT03121365/Prot_SAP_002.pdf